CLINICAL TRIAL: NCT05834647
Title: Efficacy and Safety of Prilocaine 2% and Lidocaine 5% Hyperbaric Against Spinal Anesthesia in Post Cystoscopy Procedure
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitas Sebelas Maret (Other)
Collaborators: Indonesia Endowment Fund for Education (Unknown)
Responsible Party: Principal Investigator, Septian Adi Permana. MD, Staff Department of Anesthesiology and Intensive Therapy, Universitas Sebelas Maret
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: ANES/PR/001
Record Dates: First submitted 2023-03-29; First posted 2023-04-28 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Anesthesia; Reaction; Anesthesia
Keywords: hs-CRP; Troponin; Regional Anesthesia; Cystoscopy procedure; Lidocaine; Prilocaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group P (Experimental): Drug: prilocaine 2% Dosage : 50 mg prilocaine 2% (2.5 mL volume)
  Interventions: Drug: Prilocaine 2%
- Group L (Active Comparator): Drug: hyperbaric lidocaine 5% Dosage : 50 mg hyperbaric lidocaine 5% (1 mL volume)
  Interventions: Drug: Hyperbaric Lidocaine 5%

INTERVENTIONS:
Drug: Prilocaine 2% — 50 mg prilocaine 2% (2.5 mL volume) before undergoing cystoscopy procedure
  Other Names: Takipril
  Arms: Group P
Drug: Hyperbaric Lidocaine 5% — 50 mg Hyperbaric Lidocaine 5% (1.0 mL volume) before undergoing cystoscopy procedure
  Other Names: Lidodex
  Arms: Group L

SUMMARY:
Regional anesthesia is defined as the temporary removal of nerve conduction and pain in certain areas of the body with local anesthetic drugs without causing loss of consciousness. Spinal anesthesia can provide better analgesia and shorter recovery time in urological procedures resulted in shorter operating times, lower postoperative pain, lower analgesic requirements, and shorter length of stay (LOS) compared to the general anesthesia. Lidocaine is an attractive regional anesthesia drug for ambulatory surgery since it has a rapid onset and rapid recovery from motor and sensory block. However, when it is compared with other local anesthetic agents, the use of lidocaine in spinal anesthesia is associated with an increased risk of transient neurologic symptoms, thus impeding its application to outpatient spinal anesthesia. Lidocaine is more neurotoxic than other local anesthetic agents, especially when high concentrations are applied directly to nervous tissue. Another local anesthetic agent can be used is prilocaine. It has medium potency, rapid duration, and rapid onset of action. Compared with lidocaine, prilocaine has a lower incidence of neurological symptoms in spinal anesthesia for outpatient surgery, and suitable as an alternative to long-acting low-dose local anesthetics. Therefore, the investigators intend to observe the efficacy and safety of these two agents in adult patients who will undergo cystoscopy procedure using spinal anesthesia. In this study the investigators used high-sensitivity C-Reactive Protein (hs-CRP) and high-sensitive Troponin (hs-Troponin). CRP is a systemic inflammation marker associated with conditions such as pain. Troponin can represent patient's kidney function since its metabolism and excretion are affected by changes of estimated glomerular filtration rate (eGFR). Previous study also showed that the use of spinal anesthesia can reduce the incidence of acute kidney injury. Therefore, the investigators aim to carry out further examination of the following two markers regarding to spinal anesthesia using lidocaine and prilocaine.

DETAILED DESCRIPTION:
The investigators will conduct a double-blind randomized controlled trial to compare hs-CRP and hs-Troponin levels between prilocaine 2% and hyperbaric lidocaine 5% in adult patients undergoing cystoscopy procedure with spinal anesthesia. This study was approved by the Health Research Ethics Committee (Institutional Review Board) of Dr. Moewardi General Hospital Surakarta. Before randomization, participants who are eligible based on inclusion and exclusion criteria will be given informed consent. If the patients agree, the patient will be included in this research. Ninety adult patients will be randomly divided into control group and treatment group. Control group (group L) will be given 1 mL hyperbaric lidocaine 5% (50 mg) and treatment group (group P) will be given 2.5 mL prilocaine 2% (50 mg) as spinal anesthesia. The investigators will measure hs-CRP serum levels and hs-Troponin serum levels as the primary outcome. Serum levels of hs-CRP dan hs-Troponin will be measured 4 hours postoperative.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who will undergo cystoscopy procedure with spinal anesthesia
2. Patients age between 18-60 years
3. Normal BMI according to WHO (World Health Organization) classification (18.5-24.9 kg/m2)
4. Physical status ASA (American Society of Anesthesiologists) I or ASA II according to the ASA Physical Status Classification System by the American Society of Anesthesiologists in 2020.
5. Do not have a history of disease, medication, and medical procedures related to coronary heart disease
6. There are no absolute contraindications for spinal anesthesia
7. Do not take non-steroidal analgesics and steroids within 2 weeks before surgery.
8. Do not have history and treatment of Diabetes Mellitus.
9. Willing to participate in research and sign informed consent

Exclusion Criteria:

1. Has been or will be included in other research.
2. Have a direct relative with the research team.
3. Known or suspected to HIV infection.
4. History of hypersensitivity to prilocaine or lidocaine.
5. Patients with impaired renal, hepatic, cardiac rhythm, neurologic function, myopathy, thrombocytopenia (<100,000/mL), and coagulopathy (international normalized ratio >1.5)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
hs-CRP serum level | 4 hours postoperative
  hs-CRP serum concentration will be measured using particle enhanced immunoturbidimetry method as indicator of inflammatory biomarker resulted from pain due to surgery.
hs-Troponin serum level | 4 hours postoperative
  Serum hs-Troponin at 4 hours postoperative [ Time Frame: 4 hours postoperative ] hs-Troponin serum concentration will be measured using Enzyme-Linked Fluorescent Assay (ELFA) method as indicator of kidney injury comparing lidocain 5% hyperbaric and prilocaine 2%

SECONDARY OUTCOMES:
Full regression of sensory block | Through Study Completion, an average of 1 day
  Full regression of sensory block, defined as the duration (in minutes) between intrathecal drug injection and appearance of first pain sensation reported by patients and will be confirmed by using Visual Analogue Scale. The Visual Analogue Scale (VAS) is a 10 cm or 100 mm line with anchor statements on the left scale 0 represents no pain and on the right scale 10 (or 100) represents an extreme pain. The patient is asked to mark their current pain level on the line. The examiner scores the VAS by measuring the distance in either centimeters (0 to 10) or millimeters (0 to 100) from the "no pain" anchor point.
Duration of PACU (Post-Anaesthesia Care Unit) stay | Through Study Completion, an average of 1 day
  Duration of PACU stay in minutes based on Bromage scale. Patients will be discharged from PACU if Bromage Scale <2. Bromage scale is most commonly used, although this represents only lumbosacral motor fibers and have grading scale as follow:
  0 : free movement of legs and feet with 0% blockade
  1. : just able to flex knees with free movement of feet with 33% (partial) blockade
  2. : unable to flex knee, but with free movement of feet with 66% (almost complete) blockade
  3. : unable to move legs or feet with 100% (complete) blockade
Pain score after cystoscopy procedure | Through Study Completion, an average of 1 day
  Pain score after cystoscopy procedure comparing administration of lidocaine 5% hyperbaric and prilocaine 2% using visual analogue scale (VAS) on a 100- mm VAS. The Visual Analogue Scale (VAS) is a 10 cm or 100 mm line with anchor statements on the left scale 0 represents no pain and on the right scale 10 (or 100) represents an extreme pain. The patient is asked to mark their current pain level on the line. The examiner scores the VAS by measuring the distance in either centimeters (0 to 10) or millimeters (0 to 100) from the "no pain" anchor point.
The incidence of adverse effects of hypotension | Through Study Completion, an average of 1 day
  Hypotension will be defined as a systolic blood pressure of < 90 mmHg or a decrease in mean arterial pressure (MAP in mmHg) of more than 20% from baseline preoperative value. MAP is measured from formula [(2xsystolic pressure in mmHg) + diastolic pressure in mmHg)] / 3
The incidence of adverse effects of bradycardia | Through Study Completion, an average of 1 day
  Bradycardia will be defined as heart rate < 50 beat/min
The incidence of adverse effects of nausea. | Through Study Completion, an average of 1 day
  Nausea will be assessed using (Visual Analogue Scale) VAS score for PONV (Postoperative Nausea and Vomiting). The severity of nausea was divided into four groups based on the VAS scale: 0-1 (no nausea), 1-4 (mild), 4-7 (moderate) and 7-10 (severe).

CONTACTS AND LOCATIONS:
Overall Officials: Purwoko Purwoko, PhD, Principal Investigator — Universitas Sebelas Maret

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Afari N, Mostoufi S, Noonan C, Poeschla B, Succop A, Chopko L, Strachan E. C-reactive protein and pain sensitivity: findings from female twins. Ann Behav Med. 2011 Oct;42(2):277-83. doi: 10.1007/s12160-011-9297-6. PMID 21785898
- [Result] Banerjee D, Perrett C, Banerjee A. Troponins, Acute Coronary Syndrome and Renal Disease: From Acute Kidney Injury Through End-stage Kidney Disease. Eur Cardiol. 2019 Dec 18;14(3):187-190. doi: 10.15420/ecr.2019.28.2. eCollection 2019 Dec. PMID 31933690
- [Result] Becker DE, Reed KL. Local anesthetics: review of pharmacological considerations. Anesth Prog. 2012 Summer;59(2):90-101; quiz 102-3. doi: 10.2344/0003-3006-59.2.90. PMID 22822998
- [Result] Choi HR, Song IA, Oh TK, Jeon YT. Perioperative C-reactive protein is associated with pain outcomes after major laparoscopic abdominal surgery: a retrospective analysis. J Pain Res. 2019 Mar 27;12:1041-1051. doi: 10.2147/JPR.S187249. eCollection 2019. PMID 31114292
- [Result] Ezmek B, Arslan A, Delilbasi C, Sencift K. Comparison of hemodynamic effects of lidocaine, prilocaine and mepivacaine solutions without vasoconstrictor in hypertensive patients. J Appl Oral Sci. 2010 Jul-Aug;18(4):354-9. doi: 10.1590/s1678-77572010000400006. PMID 20835569
- [Result] Garg P, Morris P, Fazlanie AL, Vijayan S, Dancso B, Dastidar AG, Plein S, Mueller C, Haaf P. Cardiac biomarkers of acute coronary syndrome: from history to high-sensitivity cardiac troponin. Intern Emerg Med. 2017 Mar;12(2):147-155. doi: 10.1007/s11739-017-1612-1. Epub 2017 Feb 11. PMID 28188579
- [Result] Hu H, Qin B, He D, Lu Y, Zhao Z, Zhang J, Wang Y, Wang S. Regional versus General Anesthesia for Percutaneous Nephrolithotomy: A Meta-Analysis. PLoS One. 2015 May 11;10(5):e0126587. doi: 10.1371/journal.pone.0126587. eCollection 2015. PMID 25961831
- [Result] Kato J, Svensson CI. Role of extracellular damage-associated molecular pattern molecules (DAMPs) as mediators of persistent pain. Prog Mol Biol Transl Sci. 2015;131:251-79. doi: 10.1016/bs.pmbts.2014.11.014. Epub 2015 Jan 30. PMID 25744676
- [Result] Koo CH, Ryu JH. Anesthetic considerations for urologic surgeries. Korean J Anesthesiol. 2020 Apr;73(2):92-102. doi: 10.4097/kja.19437. Epub 2019 Dec 17. PMID 31842248
- [Result] Manassero A, Fanelli A. Prilocaine hydrochloride 2% hyperbaric solution for intrathecal injection: a clinical review. Local Reg Anesth. 2017 Mar 31;10:15-24. doi: 10.2147/LRA.S112756. eCollection 2017. PMID 28408851
- [Result] Reece AS. High-sensitivity CRP in opiate addiction: relative and age-dependent elevations. Cardiovasc Toxicol. 2012 Jun;12(2):149-57. doi: 10.1007/s12012-012-9154-2. PMID 22297435
- [Result] Uher T, Bob P. Neuropathic pain, depressive symptoms, and C-reactive protein in sciatica patients. Int J Neurosci. 2013 Mar;123(3):204-8. doi: 10.3109/00207454.2012.746335. PMID 23126320
- [Result] Freda BJ, Tang WH, Van Lente F, Peacock WF, Francis GS. Cardiac troponins in renal insufficiency: review and clinical implications. J Am Coll Cardiol. 2002 Dec 18;40(12):2065-71. doi: 10.1016/s0735-1097(02)02608-6. PMID 12505215
- [Result] Kelley WE, Januzzi JL, Christenson RH. Increases of cardiac troponin in conditions other than acute coronary syndrome and heart failure. Clin Chem. 2009 Dec;55(12):2098-112. doi: 10.1373/clinchem.2009.130799. Epub 2009 Oct 8. PMID 19815610
- [Result] Kula A, Bansal N. Applications of cardiac biomarkers in chronic kidney disease. Curr Opin Nephrol Hypertens. 2022 Nov 1;31(6):534-540. doi: 10.1097/MNH.0000000000000829. Epub 2022 Aug 4. PMID 36004954
- See also: US National Institutes of Health, 2010. PRILOCAINE HYDROCHLORIDE injection, solution — https://dailymed.nlm.nih.gov/dailymed/drugInfo.cfm?setid=ca454f96-2e2d-46ed-95af-c741726773de
- See also: National Center for Biotechnology Information, 2022. Prilocaine — https://pubchem.ncbi.nlm.nih.gov/compound/4906